CLINICAL TRIAL: NCT07149636
Title: A Health Belief Model-Based Cross-Sectional Study on Breast Self-Examination Awareness, Practices, and Influencing Factors Among Community-Dwelling Middle-Aged and Older Women in China
Brief Title: Health Belief Model-Based Survey on Breast Self-Examination Awareness and Practice Among Community-Dwelling Middle-Aged and Older Women
Acronym: HBM-BSE
Status: Active, not recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HBM-BSE-PUMCH-2023; K8519 (Other: Peking Union Medical College Hospital Ethics Review Committee)
Record Dates: First submitted 2025-08-18; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Breast Neoplasms; Breast Self-Examination; Cancer Screening; Health Belief Model
Keywords: Breast Self-Examination; Breast Cancer Screening; Health Belief Model; Women's Health; Community Health Education; Preventive Health Behavior; Early Detection of Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Self-Examination; Health Education

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Community-Dwelling Women: Women above a certain age threshold residing in urban and suburban communities in Beijing, who meet inclusion criteria and participate in a cross-sectional survey based on the Health Belief Model regarding breast self-examination awareness and practice.

SUMMARY:
This observational study aims to evaluate the current status of breast self-examination (BSE) practices and related influencing factors among middle-aged and older women in urban communities, using the Health Belief Model (HBM) as the theoretical framework. The HBM is a well-established public health model for understanding preventive health behaviors, focusing on perceived susceptibility, perceived severity, perceived benefits, perceived barriers, cues to action, and self-efficacy.

The study will recruit community-dwelling women above approximately 40 years of age who have adequate cognitive and communication abilities. Data collection will be conducted through structured questionnaires administered during community health education activities. The survey will collect demographic information (e.g., age, occupation, education level, family history of breast cancer) and BSE-related variables, including awareness of breast cancer, perceived benefits and barriers to screening, knowledge of BSE methods, and sources of health information.

The primary outcome is the prevalence of regular BSE practices among participants. Secondary outcomes include factors associated with regular BSE performance, such as age group, occupation type, education level, family history, and knowledge of BSE techniques. Logistic regression will be used to identify independent predictors of regular BSE practices.

Findings from this study will help identify key gaps between awareness and practice, guide targeted community-based health education, and provide evidence for developing accessible, culturally appropriate breast cancer screening strategies in China. Ultimately, the results are expected to improve early detection rates and reduce the proportion of locally advanced breast cancer cases.

DETAILED DESCRIPTION:
This observational cross-sectional study is designed to investigate the prevalence and determinants of breast self-examination (BSE) practices among community-dwelling women in China, based on the Health Belief Model (HBM). Breast cancer remains the most common malignancy among women worldwide. While imaging-based screening programs have improved early detection rates in many high-income countries, large segments of the population in low- and middle-income settings still face barriers to regular breast cancer screening. In China, BSE remains a practical and low-cost complementary method for early detection, particularly in areas where mammography coverage is incomplete.

The Health Belief Model (HBM) is a theoretical framework widely used to explain preventive health behaviors and adherence to disease management. It encompasses six core dimensions: (1) perceived susceptibility to the disease, (2) perceived severity of the disease, (3) perceived benefits of preventive actions, (4) perceived barriers to taking action, (5) cues to action, and (6) self-efficacy in carrying out the preventive behavior. The present study applies the HBM framework to systematically assess the psychosocial and cognitive factors influencing BSE behaviors in Chinese women.

Study Population and Setting Participants will be recruited from multiple community health centers in Beijing. Eligible participants are women aged approximately 40 years and above, who are permanent residents in the community, possess adequate cognitive and communication abilities, and provide informed consent. Exclusion criteria include history of breast cancer, severe psychiatric illness, or inability to complete the survey.

Data Collection Procedures

Data will be collected during community health promotion activities between June 2023 and June 2025. A standardized, structured questionnaire will be used, consisting of two major sections:

1. Demographic and background information: age, occupation, education level, family history of breast cancer, and health examination history.
2. HBM-based measurement items:

   * Awareness of breast cancer as a common malignancy
   * Awareness of the importance of breast cancer screening and BSE
   * Frequency of undergoing health examinations
   * Main barriers to regular health examinations (e.g., financial concerns, lack of companion, perceived lack of necessity, other)
   * Knowledge of BSE methods and sources of information (traditional media, modern media, in-person health education)
   * Confidence in performing BSE correctly and regularly

For categorical questions, binary or multiple-choice options will be used. Open-ended questions will be coded into predefined categories based on pilot survey responses.

Quality Control Measures Prior to the study, a detailed implementation protocol and investigator manual will be developed. A pilot survey will be conducted to refine question wording and improve comprehension. During the survey, trained interviewers will strictly follow standardized procedures, avoid leading questions, and provide neutral clarifications for respondents with low literacy levels. At the end of each survey day, data will be reviewed for completeness and consistency, and invalid questionnaires will be excluded. Data entry will follow a double-entry protocol with logical checks to ensure accuracy.

Data Analysis Plan Descriptive statistics will be used to summarize demographic variables and BSE-related indicators. Categorical variables will be expressed as frequencies and percentages, and compared using Chi-square tests. Continuous variables will be expressed as mean ± standard deviation (SD) and compared using t-tests. Univariate analysis will be followed by multivariate logistic regression to identify independent predictors of regular BSE practices, with results reported as odds ratios (OR) and 95% confidence intervals (CI). A p-value < 0.05 will be considered statistically significant.

Expected Outcomes and Significance This study will quantify the gap between awareness of BSE and actual practice, identify key psychosocial and logistical barriers to regular BSE, and explore how different HBM dimensions contribute to screening behavior. The results will inform the design of tailored community-based health education programs, emphasizing skill-based training rather than solely awareness campaigns. By providing empirical evidence on screening-related behaviors in an urban Chinese population, this research will support policymakers, clinicians, and public health educators in developing culturally adapted, cost-effective strategies for breast cancer early detection.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified females aged approximately 40 years and older.
* Permanent residents of the selected community for at least 6 months.
* Able to communicate and understand the survey questions clearly.
* Provide informed consent to participate in the study.

Exclusion Criteria:

* History of breast cancer or other serious breast diseases requiring ongoing treatment.
* Cognitive impairment, severe mental illness, or other conditions affecting the ability to answer the questionnaire.
* Temporary residents or those planning to leave the community within 6 months.
* Refusal to fill out survey.

Ages: 40 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified females (including cisgender and transgender women) aged approximately 40 years and older.
Study Population: This study will recruit community-dwelling women aged approximately 40 years and above from multiple urban and suburban residential areas in Beijing, China. Participants will be permanent residents who have lived in the community for at least 6 months and are able to communicate effectively to complete the survey. The study population represents a diverse range of educational backgrounds, occupations, and health awareness levels. All participants will be enrolled during community-based health education and screening activities, and informed consent will be obtained prior to participation.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Performing Regular Breast Self-Examination (BSE) | Day 1
  Percentage of surveyed women who report performing BSE at least once per month, assessed through a standardized questionnaire at the time of study participation.

SECONDARY OUTCOMES:
Percentage of Participants Knowing the Correct Method of BSE | Day 1
  Percentage of surveyed women who report knowing how to correctly perform BSE, assessed through a structured questionnaire.
Percentage of Participants Aware of the Importance of BSE | Day 1
  Percentage of surveyed women who acknowledge the importance and health benefits of BSE, based on responses to a structured questionnaire.
Distribution of Self-Reported Barriers to Regular Health Examinations | Day 1
  Distribution of self-reported barriers to participating in regular health examinations (e.g., financial burden, lack of convenience, perceived irrelevance), assessed through a structured questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the study results will be made available to qualified researchers upon reasonable request, after publication of the primary results, for a period of 3 years. Requests will be reviewed by the study principal investigator and require a data access agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Start Date:
  6 months after publication of the primary manuscript.
  End Date:
  Available for 3 years after publication.
Access Criteria: Qualified researchers affiliated with academic or non-profit institutions may request access to the de-identified individual participant data (IPD) and supporting documents (study protocol, statistical analysis plan, informed consent form, and analytic code) for purposes of conducting scientifically valid analyses. Requests must include a research proposal outlining objectives, methodology, and intended use of the data, and will be reviewed by the study steering committee. Approved requestors will be required to sign a data sharing agreement and comply with applicable data protection regulations. Data will be shared through a secure, password-protected data repository.